CLINICAL TRIAL: NCT01391299
Title: A Multi-Centre, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Single Treatment Cycle Study of BOTOX® Cosmetic (Botulinum Toxin Type A) Purified Neurotoxin Complex in Subjects With Forehead and Glabellar Rhytides
Brief Title: Safety and Efficacy Study of Botulinum Toxin Type A for the Treatment of Forehead and Frown Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GMA-BTXC-10-002
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Facial Rhytides; Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- botulinum toxin Type A (40 Units) (Active Comparator): Botulinum toxin Type A 40 Units (total dose) injected into bilateral forehead and frown line areas on Day 1.
  Interventions: Biological: botulinum toxin Type A
- botulinum toxin Type A (30 Units) (Active Comparator): Botulinum toxin Type A 30 Units (total dose) injected into bilateral forehead and frown line areas on Day 1.
  Interventions: Biological: botulinum toxin Type A
- placebo (Normal saline) (Placebo Comparator): Placebo (Normal saline) injected into bilateral forehead and frown line areas on Day 1.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A (total dose 30 Units or 40 Units) injected into bilateral forehead and frown line areas on Day 1.
  Other Names: BOTOX® Cosmetic
  Arms: botulinum toxin Type A (30 Units); botulinum toxin Type A (40 Units)
Drug: Normal Saline — Normal Saline (placebo) injected into bilateral forehead and frown line areas on Day 1.
  Arms: placebo (Normal saline)

SUMMARY:
This study evaluated the safety and efficacy of botulinum toxin Type A compared to placebo for the treatment of forehead lines (facial rhytides) when also administered to frown lines (glabellar rhytides).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe forehead lines

Exclusion Criteria:

* Current or previous botulinum toxin treatment of any serotype within one year
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis
* Prior facial cosmetic surgery (e.g. prior periorbital surgery, facial lift, brow lift, eyelid lift or eyebrow surgery)
* Facial laser or light treatment, microdermabrasion, or superficial peels within 3 months
* Oral retinoid therapy within one year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2011-10-18 (Actual); Study Completion 2012-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Toronto, Ontario, Canada

REFERENCES:
- [Background] Solish N, Rivers JK, Humphrey S, Muhn C, Somogyi C, Lei X, Bhogal M, Caulkins C. Efficacy and Safety of OnabotulinumtoxinA Treatment of Forehead Lines: A Multicenter, Randomized, Dose-Ranging Controlled Trial. Dermatol Surg. 2016 Mar;42(3):410-9. doi: 10.1097/DSS.0000000000000626. PMID 26863598

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Normal Saline): Placebo (Normal saline) injected into bilateral forehead and frown lines areas on Day 1.
Period: Overall Study
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline)
Started | 57 | 60 | 58
Completed | 57 | 59 | 56
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 57 | 60 | 58 | 175
Age, Customized [Number; unit: Participants]
  <45 years | 28 | 25 | 22 | 75
  45 to 65 years | 26 | 31 | 35 | 92
  >65 years | 3 | 4 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 52 | 152
  Male | 7 | 10 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Score of None or Mild by Investigator-Assessed Facial Wrinkle Scale With Photonumeric Guide (FWS) in Forehead Lines at Maximum Eyebrow Elevation
Description: The Investigator assessed the severity of the patient's forehead lines at maximum eyebrow elevation using the 4-point FWS: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30.
Time Frame: Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline)
Number analyzed (Participants) | 57 | 60 | 58
Percentage of participants | 89.5 | 85.0 | 3.4

2. Primary Outcome: Percentage of Participants Achieving a Score of None or Mild by Subject-Assessed Facial Wrinkle Scale With Photonumeric Guide (FWS) in Forehead Lines at Maximum Eyebrow Elevation
Description: The patient assessed the severity of their forehead lines at maximum eyebrow elevation using the 4-point FWS: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30.
Time Frame: Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline)
Number analyzed (Participants) | 57 | 60 | 58
Percentage of participants | 87.7 | 80.0 | 6.9

3. Secondary Outcome: Percentage of Participants Achieving Satisfied or Very Satisfied by Subject Assessment of Satisfaction of Appearance of Forehead Lines
Description: Participants rated their overall satisfaction with the appearance of the forehead line area using a 5-point scale: 1=very unsatisfied, 2=unsatisfied, 3=neutral, 4=satisfied or 5=very satisfied. The percentage of participants with a rating of satisfied or very satisfied at Day 30.
Time Frame: Day 30
Population: Includes participants from the Intent-to-treat Population (all randomized participants) with a rating of very unsatisfied, unsatisfied or neutral in the Subject's Assessment of Satisfaction of Appearance at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline)
Number analyzed (Participants) | 54 | 58 | 57
Percentage of participants | 94.4 | 81.0 | 1.8

4. Secondary Outcome: Percentage of Participants With a ≥1 Grade Improvement From Baseline by Investigator-Assessed FWS in Forehead Lines at Rest
Description: The Investigator assessed the severity of the patient's forehead lines at rest using the 4-point FWS: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a ≥1 grade improvement from baseline.
Time Frame: Baseline, Day 30
Population: Participants from the intent-to-treat population (all randomized participants) with a Facial Wrinkle Score of at least mild at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline)
Number analyzed (Participants) | 56 | 60 | 58
Percentage of participants | 91.1 | 83.3 | 15.5

5. Secondary Outcome: Percentage of Participants With a ≥1 Grade Improvement From Baseline by Subject-Assessed FWS in Forehead Lines at Rest
Description: Participants assessed the severity of their forehead lines at rest using the 4-point FWS: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a ≥1 grade improvement from baseline.
Time Frame: Baseline, Day 30
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline)
Number analyzed (Participants) | 57 | 60 | 58
Percentage of participants | 89.5 | 88.3 | 17.2

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A (40 Units) | Botulinum Toxin Type A (30 Units) | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/60 | 1/58
Other Adverse Events (participants affected / at risk) | 2/57 | 8/60 | 8/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (40 Units) (N=57) | Botulinum Toxin Type A (30 Units) (N=60) | Placebo (Normal Saline) (N=58)
Nerve compression (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (40 Units) (N=57) | Botulinum Toxin Type A (30 Units) (N=60) | Placebo (Normal Saline) (N=58)
Nasopharyngitis (Infections and infestations) | 1 | 5 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Headache (Nervous system disorders) | 1 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.